CLINICAL TRIAL: NCT02909556
Title: ACURATE Neo™ AS Aortic Bioprosthesis for Implantation Using the ACURATE neoTM AS TF Transfemoral Delivery System in Patients With Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter Aortic Valve Replacement; TAVI; Transcatheter Aortic Valve Implant; Transfemoral access
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACURATE neo AS (Experimental)
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement via transfemoral access
  Other Names: ACURATE neo™ AS Aortic Bioprosthesis (Commercial name: ACURATE neo2™ Aortic Valve); ACURATE neo™ AS TF Transfemoral Delivery System (Commercial name: ACURATE neo2™ Transfemoral Delivery System)

SUMMARY:
Clinical trial aimed at evaluating the safety and performance of the ACURATE neo™ AS Aortic Bioprosthesis and ACURATE neo™ AS TF Transfemoral Delivery System for CE mark approval purposes.

DETAILED DESCRIPTION:
Single arm, prospecitve, multicenter, non-randomized and open trial. The purpose of this trial is to collect and safety and performance data concerning the ACURATE neo™ AS Aortic Bioprosthesis and ACURATE neo™ AS TF Transfemoral Delivery System

The ACURATE neo™ AS Aortic Bioprosthesis and ACURATE neo™ AS TF Transfemoral Delivery System are intended for use in minimally invasive, transcatheter aortic valve replacement (TAVR) using transfemoral access in patients presenting with severe aortic valve stenosis.

The primary objective is to evaluate the safety and performance of the study device in patients presenting with severe aortic stenosis (AS) considered to be high risk for surgery.

The secondary objective is to evaluate adverse events and study device performance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 75 years of age and older
2. Severe aortic stenosis defined as:

   * Mean aortic gradient > 40 mmHg or
   * Peak jet velocity > 4.0 m/s or
   * Aortic valve area of < 1.0 cm2
3. High risk candidate for conventional AVR defined as:

   * Logistic EuroSCORE 1 ≥ 20% or
   * STS Score ≥ 8% or
   * Heart team (cardiologist and cardiac surgeon) consensus that patient is not a surgical candidate for conventional AVR due to significant co-morbid conditions unrelated to aortic stenosis
4. NYHA Functional Class > II
5. Aortic annulus diameter from ≥ 21mm up to ≤ 27mm by CT
6. Patient willing to participate in the study and provides signed informed consent

Exclusion Criteria:

1. Congenital aortic stenosis or unicuspid or bicuspid aortic valve
2. Non-stenotic Aortic Insufficiency
3. Severe eccentricity of calcification
4. Severe mitral regurgitation (>2+)
5. Presence of mitral bioprosthesis
6. Presence of previously implanted aortic bioprosthesis
7. Presence of prosthetic ring
8. Anatomy NOT appropriate for transfemoral implant due to the size, disease and degree of calcification or tortuosity of the aorta or ilio-femoral arteries
9. Thoracic (TAA) or abdominal (AAA) aortic aneurysm
10. Presence of endovascular stent graft for treatment of TAA or AAA
11. Trans-oesophageal echocardiogram (TEE) is contraindicated
12. Evidence of intra-cardiac mass, thrombus or vegetation
13. Severe ventricular dysfunction with ejection fraction < 20%
14. Any percutaneous intervention, except for balloon valvuloplasty (BAV) within 1 month prior to implant procedure
15. Acute Myocardial Infarction within 1 month prior to implant procedure
16. Previous TIA or stroke within 3 months prior to implant procedure
17. Active ulcer or gastrointestinal (GI) bleeding within 3 months prior to implant procedure
18. Any scheduled surgical or percutaneous procedure to be performed prior to 30 day visit
19. Severe coagulation conditions
20. Refusal of blood transfusions
21. Systolic pressure <80mmHg, cardiogenic shock, need for inotropic support or IABP
22. Hypertrophic cardiomyopathy with or without obstruction
23. Active bacterial endocarditis or other active infections
24. Hepatic failure (> Child B)
25. Chronic renal dysfunction with serum creatinine > 2.5 mg/dL or renal dialysis
26. Refusal of surgery
27. Severe COPD requiring home oxygen
28. Neurological disease severely affecting ambulation or daily functioning, or dementia
29. Life expectancy < 12 months due to non-cardiac co-morbid conditions
30. Inability to tolerate anticoagulation therapy
31. Contraindication to contrast media or allergy to nickel
32. Currently participating in an investigational drug or another device study
33. Non-valvular aortic stenosis
34. Non-calcific acquired aortic stenosis

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 30 days follow-up | 30 days post-implant

SECONDARY OUTCOMES:
Rate of clinical events as defined per VARC guidelines | 7 days, 30 days, 12 months post-implant
  Clinical events:
  * Mortality
  * Stroke
  * Myocardial infarction
  * Bleeding complication
  * Acute kidney injury
  * Vascular complication
  * Conduction disturbances and arrhythmia
  * Other TAVI-related complications
Procedural success | Day of implant
  2. Procedural success defined as absence of complications arising during implantation of the prosthetic valve such as: inability to properly seat the valve in the annulus; need for more than one aortic bioprosthesis (valve in valve); or if a surgical aortic valve replacement is required to correct a severe aortic regurgitation or procedure complication
Device success | Day of implant
  3. Device success defined as:
  * Absence of intra-procedure mortality AND,
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND,
  * Intended performance of the prosthetic heart valve (EOAi >0.85 cm2/m2 and mean aortic valve gradient <20mmHg without moderate or severe AR)
VARC Composite Safety at 30 days | 30 days
Clinical improvement from baseline as per NYHA Functional Classification | 7 days, 30 days, 12 months post-implant
Improvement from baseline in hemodynamic function: effective orifice area, mean transprosthetic gradient | 7 days, 30 days, 12 months
Total aortic regurgitation | 7 days, 30 days, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helge Möllmann, Prof., Principal Investigator — Klinik für Innere Medizin - St.-Johannes-Hospital - Dortmund, Germany
Locations (9):
- Rigshospitalet, Copenhagen, Denmark
- Germany (7):
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - Johannes Hospital, Dortmund
  - Universitätsklinikum Halle - Universitätsklinik und Poliklinik für Herzchirurgie, Halle
  - Universitäres Herzzentrum Hamburg - Klinik und Poliklinik für Herz- und Gefäßchirurgie, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, München
  - Universitätsklinik Regensburg, Regensburg
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)